CLINICAL TRIAL: NCT04169178
Title: A Phase 1 Dose Finding/Expansion Study of HLX55, A Monoclonal Antibody Targeting Tyrosine-Protein Kinase MET (C-MET) in Patients With Advanced Solide Tumors Refactory to Standard Therapy
Brief Title: Evaluate Safety, Tolerability and PK of HLX55 in Patients With Advanced Solid Tumors With Different cMET Status
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henlix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLX55-001
Record Dates: First submitted 2019-11-13; First posted 2019-11-19 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HLX55, dose finding stage, advanced solid tumor (Experimental): Participants will receive HLX55 at assign dose level, e.g. 2.5, 5, 15 and 25 mg/kg every three weeks followed by a 21-day DLT observation period.
  Interventions: Drug: HLX55
- HLX55, dose expansion stage, gastric cancer (Experimental): Participants diagnosed with gastric cancer with will receive HLX55 in recommended phase 2 dose (RP2D) every three weeks.
  Interventions: Drug: HLX55
- HLX55, dose expansion stage, NSCLC (Experimental): Participants diagnosed with non-small cell lung cancer (NSCLC) with will receive HLX55 in RP2D every three weeks.
  Interventions: Drug: HLX55
- HLX55, dose expansion stage, colorectal cancer (Experimental): Participants diagnosed with colorectal cancer (CRC) with will receive HLX55 in RP2D every three weeks.
  Interventions: Drug: HLX55
- HLX55, dose expansion stage, other solid cancer (Experimental): Participants diagnosed with other solid cancer with will receive HLX55 in RP2D every three weeks.
  Interventions: Drug: HLX55

INTERVENTIONS:
Drug: HLX55 — A humanized IgG2 monoclonal antibody targeting tyrosine-protein kinase MET (c-MET)
  Other Names: HLX55 monoclonal antibody for Injection

SUMMARY:
A mutilpe-center, open-label, dose-escalation Phase I clinical trial to evaluate the safety and the tolerability of HLX55 in patients with advanced solid tumors overexpressing/Mutation/Amplification cMET after failure of standard of care.

DETAILED DESCRIPTION:
This study is an open-label and dose escalation study including dose finding stage and expansion stage.

In dosing finding stage, the study will precede in two phases, (i) a modified accelerated titration design 2A (ATD 2A) phase and (ii) a traditional 3+3 dose escalation phase aimed at exploring the safety and MTD of HLX55. Four dose levels are designed for HLX55 in this stage: 2.5, 5, 15, and 25 mg/kg/3 weeks. The 5 mg/kg/3 weeks will serve as the starting dose.

In the dose-expansion stage, three to five cohorts are planned, and different cohorts will evaluate the efficacy of HLX55 for potential indications. Maximum 20 patients will be accrued in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients must be 18-years of age or older (or per local regulations) and ≦75 years of age.
2. For dose finding stage: patients with measurable or evaluable advanced or metastatic solid tumours who have failed standard therapy or for whom no standard therapy is available.
3. For dose expansion stage: patients with measurable or evaluable advanced or metastatic solid tumors with histologically confirmed c-MET mutations (MET exon 14 mutations) or amplifications (MET/CEP7 ratio ≥ 2.0 or MET ≥ 5.0 copies) or over-expression (immunohistochemistry [IHC] score ≥ 2+) and have failed standard therapy or for whom no standard therapy is available. Positive c-MET mutation/amplification/over-expression results should be available before the subject can receive HLX55.
4. No prior therapy with MET-targeting biological agents (patients who have received prior therapy with a MET-targeting tyrosine kinase inhibitor [TKI] is allowed.)
5. Must be able to supply adequate tumor tissue. (Adequate tumor biopsy material means (1) newly biopsied or archival tissue biopsied within 60 days before the first dosing, (2) Biopsy materials should be adequate for biomarker analysis (c-MET/Kras/EGFR).
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at the time of study entry.
7. Able to provide informed consent.
8. A life expectancy longer than three months.
9. Adequate hematologic functions, as defined by absolute neutrophil counts ≥ 1500/mm3; a haemoglobin level ≥ 9 gm/dL; a platelet count ≥ 100,000/mm3 and an international normalized ratio ≤ 1.5.
10. An adequate hepatic function defined by a total bilirubin level ≤ 1.5 x of upper limit of normal values (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 2.5 x of ULN or ≤ 5 x of ULN in known hepatic metastases or with primary hepatocellular carcinoma.
11. Adequate renal function, as defined by the creatinine clearance rate ≥ 50 mL/minute by Cockcroft-Gault formula. In patients with extreme body weights (body mass index [BMI] < 18.5 OR > 30) estimated glomerular filtration rate (eGFR) ≥ 50ml/min calculated by Modification of Diet in Renal Disease (MDRD) formula is acceptable.
12. Adequate cardiac function defined as left ventricular ejection fraction (LVEF) ≥ 50% measured by either cardiac echo or multigated acquisition (MUGA) scan.
13. At least 21days from prior cytotoxic chemotherapy, prior therapy with investigational small molecule agents (or medical device) or radiotherapy, at least 28 days from prior immunotherapy, biological agents or prior major surgery and at least 14 days from prior hormonal therapy and minor surgery before infusion of first dose of HLX55.
14. For patients with hepatocellular carcinoma, their Child-Pugh score must be A.
15. Able to be followed up as required by the study protocol.
16. Female participants must have a negative pregnancy test at screening if of childbearing potential or be of non-childbearing potential.
17. Female participants of childbearing potential and male partners with female partners of childbearing potential must agree to use 2 adequate barrier methods of contraception during the study and for at least 180 days after last dose of study drug.

Exclusion Criteria:

1. Patients who still have ≥ grade 2 toxicities from prior therapies.
2. Concurrent unstable or uncontrolled medical conditions with either of the followings:

   * Active systemic infections requiring intravenous antibiotic use within 1 week;
   * Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg), or poor compliance with anti-hypertensive agents;
   * Clinically significant arrhythmia requiring anti-arrhythmia therapy, unstable angina pectoris, congestive heart failure (class III or IV of New York Heart Association [NYHA]) or acute myocardial infarction within 6 months;
   * Uncontrolled diabetes or poor compliance with hypoglycemics defined by glycated hemoglobin (HbA1c) ≥ 9.5%;
   * The presence of chronically unhealed wound or ulcers;
   * Uncontrolled hypercalcemia (defined as persistent Ionized (free) Calcium ≥ 6.5 mg/dl despite appropriate management.)
   * Other chronic diseases, which, in the opinion of the investigator, could compromise the safety of the patient or the integrity of the study.
3. Newly-diagnosed or symptomatic brain metastases (patients with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and not taking steroids for brain edema at least 14 days before infusion of the first dose of HLX55 can be allowed in the study). Anticonvulsants are allowed.
4. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 3 years can participate).
5. Known history of human immunodeficiency virus infection (HIV), hepatitis B virus carrier status (HBV surface antigen positive) and hepatitis C carrier (anti-HCV antibody positive).
6. The patient is the investigator, sub-investigator or anyone directly involved in the conduct of the study.
7. History or current evidence of any condition or disease that could confound the results of the study or, in the opinion of Investigator(s), is not in the best interest of the patient to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Dose finding stage-safety | Up to 2 years
  Numbers and percentage of patients with adverse events (AEs).
Dose finding stage-MTD or RP2D | Up to 2 years
  The maximum tolerated dose and recommended phase 2 dose (RP2D) of HLX55.
Dose expansion stage-safety | Up to 2 years
  Numbers and percentage of patients with adverse events (AEs).
Dose expansion stage-efficacy | Up to 2 years
  Disease control rate (DCR).
Dose expansion stage-efficacy | Up to 2 years
  Overall response rate (ORR).
Dose expansion stage-efficacy | Up to 2 years
  Duration of response (DOR).

SECONDARY OUTCOMES:
Dose finding stage and dose expansion stage-PK profile | Through study completion, up to 2 years.
  PK profile of HLX55 including maximum concentration (Cmax), minimum concentration (Cmin), area under concentration (AUC0-tau), half-life (T1/2), clearance (CL) rate and the volume of distribution at steady state (Vss) at different doses.
Dose finding stage and dose expansion stage-serum HGF levels | Cycle 1 to 3 (each cycle is 21 days)
  Changes in serum HGF levels before and at different time-points after HLX55 treatment.
Dose finding stage and dose expansion stage-immunogenicity | Up to 2 years
  The presence and percentage of anti-HLX55 antibody-positive patients (immunogenicity) by measurement of anti-HLX55 antibodies in serum.

OTHER OUTCOMES:
Dose finding stage and dose expansion stage-cMET status | up to 3 cycles (each cycle is 21 days)
  Relationship between levels or status of c-MET mutations/overexpression/amplification, EGFR mutation and KRAS mutation

CONTACTS AND LOCATIONS:
Overall Officials: Tsu-Yi Chao, MD. PhD., Principal Investigator — Shuang Ho Hospital,Ministry of Health and Welfare, Taipei, Taiwan; Ching-Liang Ho, MD, Principal Investigator — Tri-Service General Hospital, Taipei, Taiwan; Wu-Chou Su, MD. PhD., Principal Investigator — National Cheng Kung University Hospital, Tainan, Taiwan; Chia-Lun Chang, MD, Principal Investigator — Taipei Municipal Wanfang Hospital, Taipei, Taiwan
Locations (4):
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - Tri-Service General Hospital, Taipei
  - Taipei Minicipal Wangfang Hospital, Taipei
  - Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, Taipei County

IPD SHARING:
Plan to Share IPD: No